CLINICAL TRIAL: NCT07172386
Title: A Study on the Safety and Efficacy of Super-selective Tumour Arterial Embolisation in Combination With Toripalimab and Axitinib as a Preoperative Treatment for Advanced Renal Cell Carcinoma
Brief Title: Preoperative Therapy of Super-selective Tumor Artery Embolization Combined With Toripalimab and Axitinib in Advanced RCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SETAR
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Renal Cell Carcinoma (RCC)
Keywords: Toripalimab; Axitinib; Super-selective renal artery embolization; Advanced Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — toripalimab; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Embolization plus toripalimab and axitinib (Experimental): Patients will undergo super-selective embolization of the feeding arteries to the renal tumour one week prior to drug therapy, followed by toripalimab administered every three weeks for four consecutive cycles combined with axitinib administered for four consecutive cycles in the preoperative and patients need to continue taking the drug for a year after surgery
  Interventions: Drug: Toripalimab and axitinib

INTERVENTIONS:
Drug: Toripalimab and axitinib — Patients will undergo super-selective embolization of the feeding arteries to the renal tumour one week prior to drug therapy, followed by toripalimab administered every three weeks for four consecutive cycles combined with axitinib administered for four consecutive cycles before surgery, and followed by 17 cycles' toripalimab for adjuvant therapy.
  Other Names: Super-selective tumor arterial embolization

SUMMARY:
This is a phase II study to determine the efficacy and safety of Super-selective tumor artery embolization combined with toripalimab and axitinib as treatment for patients with the advanced kidney cancer . Further evaluate whether the treatment plan is beneficial to the patient's operation. Patients will undergo super-selective embolization of the feeding arteries to the renal tumour one week prior to drug therapy, followed by toripalimab administered every three weeks for three to four consecutive cycles combined with axitinib administered for four consecutive cycles in the preoperative and patients need to continue taking the drug for a year after surgery

DETAILED DESCRIPTION:
This is a phase II study to determine the efficacy and safety of Super-selective tumor artery embolization combined with toripalimab and axitinib as treatment for patients with the advanced kidney cancer . Further evaluate whether the treatment plan is beneficial to the patient's operation. Patients will undergo super-selective embolization of the feeding arteries to the renal tumour one week prior to drug therapy, followed by toripalimab administered every three weeks for three to four consecutive cycles combined with axitinib administered for four consecutive cycles in the preoperative and patients need to continue taking the drug for a year after surgery, The main objective of the study was to evaluate whether the treatment was beneficial to patients undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Age ≥ 18 years
* Patients with pathologically and radiographically confirmed renal cell carcinoma:

  * cT2N0M0 with Grade 4 or sarcomatoid feature;
  * cT3-4N0M0;
  * cTanyN1M0;
  * M1 that can be returned to M0 through local therapy
* Preoperative imaging evaluation can be performed radical excision or tumor reduction surgery
* There are no suspected brain metastases
* The presence of measurable lesions was assessed according to RECISTv1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Organ function level must meet the following requirements: Hematological indexes: neutrophil count >= 1.5x10^9/L, platelet count >= 100x10^9/L, hemoglobin >= 9.0 g/dl (can be maintained by blood transfusion); Liver function: total bilirubin <=1.5 ULN, alanine aminotransferase and aspartate aminotransferase <=1.5 ULN
* Non-surgically sterilized or reproductive-age female patients must use a medically approved contraceptive method (such as an intrauterine device, oral contraceptives, or condoms) during the study treatment period and for 3 months after its completion; Female patients who are not surgically sterilized or are of childbearing potential must have a negative serum or urine HCG test within 7 days prior to study enrollment and must not be lactating. Male patients who are not surgically sterilized or are of childbearing potential must agree to use one medically approved contraceptive method with their spouse during the study treatment period and for 3 months after the study treatment period ends.
* The subjects volunteered to join the study, signed informed consent, and had good compliance with follow-up

Exclusion Criteria:

* Prior receipt of radiotherapy, chemotherapy, long-term or high-dose corticosteroid therapy, surgery, or molecular targeted therapy
* Subjects with a history of or concurrent other malignancies (except those controllable and not affecting 2-year survival)
* Prior treatment with other PD-1/PD-L1 therapies; Known history of allergy to macromolecular protein preparations or any known PD-1 component
* Active autoimmune disease or history of autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; Subjects with vitiligo or childhood asthma that has achieved complete remission without requiring any intervention in adulthood may be included; subjects requiring medical intervention with bronchodilators for asthma are excluded);
* Subjects currently using immunosuppressive agents for immunosuppression purposes and continuing such use within 2 weeks prior to enrollment
* Uncontrolled cardiac clinical symptoms or diseases, such as:

  * New York Heart Association (NYHA) Class II or higher heart failure;
  * Unstable angina;
  * Myocardial infarction within the past year;
  * Clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention
* Coagulation abnormalities (PT > 16s, APTT > 43s, TT > 21s, Fbg > 2g/L) with bleeding tendency or currently receiving thrombolytic or anticoagulant therapy;
* Active gastrointestinal bleeding within 3 months prior to first dose due to esophageal varices, active gastric or duodenal ulcer, ulcerative colitis, portal hypertension, or unresected tumors; or other conditions judged by the investigator to potentially cause gastrointestinal bleeding or perforation
* History or current presence of major bleeding (≥30 mL within 3 months), hemoptysis (≥5 mL fresh blood within 4 weeks), or thromboembolic events (including stroke and/or transient ischemic attack) within 12 months
* Active infection or unexplained fever >38.5°C occurring during screening or prior to first dose
* History of abdominal fistula, gastrointestinal perforation, or abdominal abscess within 4 weeks prior to first dose
* Objective evidence of past or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, or severe pulmonary impairment
* Subjects with congenital or acquired immunodeficiency, such as HIV infection, or active hepatitis (transaminase levels not meeting inclusion criteria; for hepatitis B: HBV DNA ≥10⁴/ml; for hepatitis C: HCV RNA ≥10³/ml); chronic hepatitis B virus carriers with HBV DNA ≥2000 IU/ml (≥10⁴ copies/ml) must concurrently receive antiviral therapy during the study to be eligible for enrollment
* Subjects currently participating in other clinical studies or those who completed a prior clinical study within the past month; subjects may receive other systemic antitumor therapies during the study period
* Administration of live vaccines within 4 weeks prior to study drug initiation or during the study period
* Known history of psychiatric drug abuse, alcoholism, or substance abuse;
* Inability or refusal to bear out-of-pocket costs for examinations and treatments
* The investigator deems the subject should be excluded from this study, such as when the investigator determines the subject has other factors that may necessitate premature termination of the study, including: other serious illnesses (including psychiatric disorders) requiring concomitant treatment, severe laboratory abnormalities, or family/social factors that may compromise subject safety or interfere with data/sample collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
R0 Resection Rate | through study completion, an average of 3 year
  The proportion of patients who achieve complete resection with no residual tumor cells detected at the surgical margin, serving as a primary outcome measure to assess the success of surgical intervention in the study.
ORR | through study completion, an average of 3 year
  According to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, the objective response rate (ORR) following preoperative treatment was assessed by the investigator.
Preoperative Treatment Safety: Treatment-Related Side Effects | Through treatment completion (before surgery), an average of 4 cycles (each cycle is 21 days)
  Treatment-Related Side Effects

SECONDARY OUTCOMES:
Perioperative Complications | Throughout treatment until 30 days after surgery
  Intraoperative Blood Loss, Karnofsky Score, and Hospital Stay
Progression free survival | Every 12 weeks until 12 months after surgery
  Progression free survival was assessed by imaging (enhanced CT, enhanced MRI or both ) after surgery every 12 weeks until 12 months.
Major Pathological Response | Within 14 days after surgical resection
  Defined as ≤10% residual viable tumor cells in the resected tumor specimen (assessed by pathological examination after surgery). Serves as a secondary outcome to evaluate the effectiveness of preoperative therapy in reducing tumor burden at the pathological level.
Patient-Reported Quality of Life | Through adjuvant treatment completion (after surgery), with assessments once every 3 weeks for a total of 17 cycles (each cycle is 21 days)
  EORTC QLQ-C30 and FKSI-15 Scores
Overall Survival (OS) | Follow-up is performed once every 3 months (±14 days)
  Subjects will undergo survival follow-up until the earliest occurrence of the following events: subject death, loss to follow-up, withdrawal of informed consent, completion of 5 years of survival follow-up, or study termination.

OTHER OUTCOMES:
Rate of responser with predictive biomarker positive | Through treatment completion (before surgery), an average of 4 cycles (each cycle is 21 days)
  Bulk RNA-seq and/or single cell RNA-seq were performed in part of tissues before and after neoadjuvant treatment to seek biomarkers predicting Response

CONTACTS AND LOCATIONS:
Overall Officials: Changyi Quan, MD, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical University Second Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Background] ournal/Source：Presented at: American Society of Clinical Oncology - Genitourinary Cancers Symposium (ASCO - GU) 2025 • Publication Year：2025 • Other Info：Abstract #477684
- [Background] Muller A, Rouviere O. Renal artery embolization-indications, technical approaches and outcomes. Nat Rev Nephrol. 2015 May;11(5):288-301. doi: 10.1038/nrneph.2014.231. Epub 2014 Dec 23. PMID 25536394
- [Background] Rothrock NE, Jensen SE, Beaumont JL, Abernethy AP, Jacobsen PB, Syrjala K, Cella D. Development and initial validation of the NCCN/FACT symptom index for advanced kidney cancer. Value Health. 2013 Jul-Aug;16(5):789-96. doi: 10.1016/j.jval.2013.04.015. Epub 2013 Jun 19. PMID 23947972
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Powles T, Plimack ER, Soulieres D, Waddell T, Stus V, Gafanov R, Nosov D, Pouliot F, Melichar B, Vynnychenko I, Azevedo SJ, Borchiellini D, McDermott RS, Bedke J, Tamada S, Yin L, Chen M, Molife LR, Atkins MB, Rini BI. Pembrolizumab plus axitinib versus sunitinib monotherapy as first-line treatment of advanced renal cell carcinoma (KEYNOTE-426): extended follow-up from a randomised, open-label, phase 3 trial. Lancet Oncol. 2020 Dec;21(12):1563-1573. doi: 10.1016/S1470-2045(20)30436-8. Epub 2020 Oct 23. PMID 33284113
- [Background] Motzer RJ, Hutson TE, Cella D, Reeves J, Hawkins R, Guo J, Nathan P, Staehler M, de Souza P, Merchan JR, Boleti E, Fife K, Jin J, Jones R, Uemura H, De Giorgi U, Harmenberg U, Wang J, Sternberg CN, Deen K, McCann L, Hackshaw MD, Crescenzo R, Pandite LN, Choueiri TK. Pazopanib versus sunitinib in metastatic renal-cell carcinoma. N Engl J Med. 2013 Aug 22;369(8):722-31. doi: 10.1056/NEJMoa1303989. PMID 23964934
- [Background] Motzer RJ, Tannir NM, McDermott DF, Aren Frontera O, Melichar B, Choueiri TK, Plimack ER, Barthelemy P, Porta C, George S, Powles T, Donskov F, Neiman V, Kollmannsberger CK, Salman P, Gurney H, Hawkins R, Ravaud A, Grimm MO, Bracarda S, Barrios CH, Tomita Y, Castellano D, Rini BI, Chen AC, Mekan S, McHenry MB, Wind-Rotolo M, Doan J, Sharma P, Hammers HJ, Escudier B; CheckMate 214 Investigators. Nivolumab plus Ipilimumab versus Sunitinib in Advanced Renal-Cell Carcinoma. N Engl J Med. 2018 Apr 5;378(14):1277-1290. doi: 10.1056/NEJMoa1712126. Epub 2018 Mar 21. PMID 29562145
- [Background] Zhang Z, Xiong L, Wu Z, Liu H, Ning K, Peng Y, Yu C, Ding Y, Weng D, Xia J, Jiang L, Guo S, Han H, Zhou F, Dong P. Neoadjuvant combination of pazopanib or axitinib and programmed cell death protein-1-activated dendritic cell-cytokine-induced killer cells immunotherapy may facilitate surgery in patients with renal cell carcinoma. Transl Androl Urol. 2021 May;10(5):2091-2102. doi: 10.21037/tau-21-406. PMID 34159090
- [Background] Liu J, Blake SJ, Yong MC, Harjunpaa H, Ngiow SF, Takeda K, Young A, O'Donnell JS, Allen S, Smyth MJ, Teng MW. Improved Efficacy of Neoadjuvant Compared to Adjuvant Immunotherapy to Eradicate Metastatic Disease. Cancer Discov. 2016 Dec;6(12):1382-1399. doi: 10.1158/2159-8290.CD-16-0577. Epub 2016 Sep 23. PMID 27663893
- [Background] Gorin MA, Patel HD, Rowe SP, Hahn NM, Hammers HJ, Pons A, Trock BJ, Pierorazio PM, Nirschl TR, Salles DC, Stein JE, Lotan TL, Taube JM, Drake CG, Allaf ME. Neoadjuvant Nivolumab in Patients with High-risk Nonmetastatic Renal Cell Carcinoma. Eur Urol Oncol. 2022 Feb;5(1):113-117. doi: 10.1016/j.euo.2021.04.002. Epub 2021 May 26. PMID 34049847
- [Background] Chapin BF, Delacroix SE Jr, Culp SH, Nogueras Gonzalez GM, Tannir NM, Jonasch E, Tamboli P, Wood CG. Safety of presurgical targeted therapy in the setting of metastatic renal cell carcinoma. Eur Urol. 2011 Nov;60(5):964-71. doi: 10.1016/j.eururo.2011.05.032. Epub 2011 May 25. PMID 21621907
- [Background] Borregales LD, Adibi M, Thomas AZ, Wood CG, Karam JA. The role of neoadjuvant therapy in the management of locally advanced renal cell carcinoma. Ther Adv Urol. 2016 Apr;8(2):130-41. doi: 10.1177/1756287215612962. Epub 2015 Nov 20. PMID 27034725
- [Background] Motzer RJ, Ravaud A, Patard JJ, Pandha HS, George DJ, Patel A, Chang YH, Escudier B, Donskov F, Magheli A, Carteni G, Laguerre B, Tomczak P, Breza J, Gerletti P, Lechuga M, Lin X, Casey M, Serfass L, Pantuck AJ, Staehler M. Adjuvant Sunitinib for High-risk Renal Cell Carcinoma After Nephrectomy: Subgroup Analyses and Updated Overall Survival Results. Eur Urol. 2018 Jan;73(1):62-68. doi: 10.1016/j.eururo.2017.09.008. Epub 2017 Sep 28. PMID 28967554
- [Background] Gross-Goupil M, Kwon TG, Eto M, Ye D, Miyake H, Seo SI, Byun SS, Lee JL, Master V, Jin J, DeBenedetto R, Linke R, Casey M, Rosbrook B, Lechuga M, Valota O, Grande E, Quinn DI. Axitinib versus placebo as an adjuvant treatment of renal cell carcinoma: results from the phase III, randomized ATLAS trial. Ann Oncol. 2018 Dec 1;29(12):2371-2378. doi: 10.1093/annonc/mdy454. PMID 30346481
- [Background] Motzer RJ, Haas NB, Donskov F, Gross-Goupil M, Varlamov S, Kopyltsov E, Lee JL, Melichar B, Rini BI, Choueiri TK, Zemanova M, Wood LA, Reaume MN, Stenzl A, Chowdhury S, Lim HY, McDermott R, Michael A, Bao W, Carrasco-Alfonso MJ, Aimone P, Voi M, Doehn C, Russo P, Sternberg CN; PROTECT investigators. Randomized Phase III Trial of Adjuvant Pazopanib Versus Placebo After Nephrectomy in Patients With Localized or Locally Advanced Renal Cell Carcinoma. J Clin Oncol. 2017 Dec 10;35(35):3916-3923. doi: 10.1200/JCO.2017.73.5324. Epub 2017 Sep 13. PMID 28902533
- [Background] Haas NB, Manola J, Uzzo RG, Flaherty KT, Wood CG, Kane C, Jewett M, Dutcher JP, Atkins MB, Pins M, Wilding G, Cella D, Wagner L, Matin S, Kuzel TM, Sexton WJ, Wong YN, Choueiri TK, Pili R, Puzanov I, Kohli M, Stadler W, Carducci M, Coomes R, DiPaola RS. Adjuvant sunitinib or sorafenib for high-risk, non-metastatic renal-cell carcinoma (ECOG-ACRIN E2805): a double-blind, placebo-controlled, randomised, phase 3 trial. Lancet. 2016 May 14;387(10032):2008-16. doi: 10.1016/S0140-6736(16)00559-6. Epub 2016 Mar 9. PMID 26969090
- [Background] Ravaud A, Motzer RJ, Pandha HS, George DJ, Pantuck AJ, Patel A, Chang YH, Escudier B, Donskov F, Magheli A, Carteni G, Laguerre B, Tomczak P, Breza J, Gerletti P, Lechuga M, Lin X, Martini JF, Ramaswamy K, Casey M, Staehler M, Patard JJ; S-TRAC Investigators. Adjuvant Sunitinib in High-Risk Renal-Cell Carcinoma after Nephrectomy. N Engl J Med. 2016 Dec 8;375(23):2246-2254. doi: 10.1056/NEJMoa1611406. Epub 2016 Oct 9. PMID 27718781
- [Background] Choueiri TK, Tomczak P, Park SH, Venugopal B, Ferguson T, Chang YH, Hajek J, Symeonides SN, Lee JL, Sarwar N, Thiery-Vuillemin A, Gross-Goupil M, Mahave M, Haas NB, Sawrycki P, Gurney H, Chevreau C, Melichar B, Kopyltsov E, Alva A, Burke JM, Doshi G, Topart D, Oudard S, Hammers H, Kitamura H, Bedke J, Perini RF, Zhang P, Imai K, Willemann-Rogerio J, Quinn DI, Powles T; KEYNOTE-564 Investigators. Adjuvant Pembrolizumab after Nephrectomy in Renal-Cell Carcinoma. N Engl J Med. 2021 Aug 19;385(8):683-694. doi: 10.1056/NEJMoa2106391. PMID 34407342
- [Background] Speed JM, Trinh QD, Choueiri TK, Sun M. Recurrence in Localized Renal Cell Carcinoma: a Systematic Review of Contemporary Data. Curr Urol Rep. 2017 Feb;18(2):15. doi: 10.1007/s11934-017-0661-3. PMID 28213859